CLINICAL TRIAL: NCT00042445
Title: Brain Neoplasms, Leukemia and Petrochemical Exposures
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Collaborators: Harvard School of Public Health (HSPH) (Other); Kaohsiung Medical University (Other)
Other Study IDs: 9723-CP-001
Record Dates: First submitted 2002-07-30; First posted 2002-08-01 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Leukemia; Brain Neoplasm
Keywords: Neoplasm; Petrochemical; Leukemia; Taiwan
MeSH Terms: conditions — Leukemia; Brain Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control

SUMMARY:
The aim of this study is to examine the association of exposure to air contaminants (PAH & VOC) emitted from the petrochemical industries, specific genetic polymorphisms (P4501A1 (MspI & exon 7) and GSTM1 & T1) of study subjects and their parents, and the risks of brain tumors and leukemia among children and youths in metropolitan Kaohsiung, southern Taiwan.

DETAILED DESCRIPTION:
Brain tumors and leukemia are the most common malignancies among children and adolescents in the U.S. Adequate information on the role of inherited genetic susceptibility and environmental exposures in the development of neoplasms in children and adolescents is lacking. In Taiwan, four large petrochemical industries are located in the Kaohsiung metropolitan area. These facilities are proximal to residential areas because of the high population density in the region. Data have shown that the concentrations of ambient polycyclic aromatic hydrocarbons (PAH) and volatile organic compounds (VOC) around the petrochemical industries are at least 10 and 2 times, respectively, higher than those in U.S. industrialized communities. Our preliminary case-control study in metropolitan Kaohsiung showed that young residents (under age 30) living within 3 kilometers of the vicinity of petrochemical industries have a 6.0 fold increase in brain neoplasms and a 2.9 fold increase in leukemia. The purpose of this proposal is to examine the association of exposure to air contaminants (PAH and VOC) emitted from the petrochemical industries, specific genetic polymorphisms (P4501A1 (MspI & exon 7) and GSTM1 &T1) from study subjects and their parents, and the risks of brain tumors and leukemia among children and youths in metropolitan Kaohsiung. Our hypothesis is that there is an increased risk of brain tumors and leukemia in patients with high cumulative exposure to these hazards, and that heritable polymorphisms in several genes modify this association. In addition to an independent association of environmental and genetic factors with brain neoplasms and leukemia, we hypothesize that there is greater risk associated with the presence of combined environmental exposure and the high risk genotype. Also, we will assess the role of parental genetic polymorphisms in the development of cancer in their siblings. This proposed study uses an environmental molecular epidemiologic approach, utilizing prospective enrollment of a cohort of brain tumor and leukemia subjects in a population-based case-control design. This proposal is responsive to the recommendation of the National Research Council that risk assessment and public health policy pay special attention to the protection of children.

ELIGIBILITY:
Young population Less than 30 Resident of Kaohsiung metropolitan, Taiwan

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1456
Dates: Start 2000-08; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Locations (2):
- Harvard School of Public Health, Boston, Massachusetts, United States
- Kaohsiung Medical University, Kaohsiung City, Taiwan